CLINICAL TRIAL: NCT03112941
Title: Hyperbaric Oxygen and Orthopedic Comprehensive Treatment for Traumatic Incomplete Spinal Cord Injury in the Plateau: an Open-label Randomized Controlled Clinical Trial
Brief Title: Hyperbaric Oxygen and Orthopedic Comprehensive Treatment for Traumatic Incomplete Spinal Cord Injury in the Plateau
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Jun Ma, Principal Investigator, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_JM
Record Dates: First submitted 2017-04-08; First posted 2017-04-13 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 164 patients with traumatic incomplete spinal cord injury (SCI) were recruited in the plateau from June 2012 to February 2016.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Patients with traumatic incomplete spinal cord injury (SCI) in the control group are treated with pedicle screw fixation and decompressive laminectomy.
  Interventions: Procedure: control group
- hyperbaric oxygen group (Experimental): Patients with traumatic incomplete spinal cord injury (SCI) in the hyperbaric oxygen group are treated with pedicle screw fixation and decompressive laminectomy, and are given 0.2 MPa hyperbaric oxygen (HBO), once a day, 10 times as a course, with 5-7 days of resting between two courses, totally four courses.
  Interventions: Other: hyperbaric oxygen group

INTERVENTIONS:
Procedure: control group — Patients with traumatic incomplete spinal cord injury (SCI) in the control group are treated with pedicle screw fixation and decompressive laminectomy.
  Arms: control group
Other: hyperbaric oxygen group — Patients with traumatic incomplete spinal cord injury (SCI) in the hyperbaric oxygen group are treated with pedicle screw fixation and decompressive laminectomy, and are given 0.2 MPa hyperbaric oxygen (HBO), once a day, 10 times as a course, with 5-7 days of resting between two courses, totally four courses.
  Arms: hyperbaric oxygen group

SUMMARY:
To observe modified Barthel index, American Spinal Injury Association (ASIA) impairment scale grading, sensory score and motor score in patients with incomplete SCI in the plateau using 0.2 MPa HBO combined with pedicle screw fixation and decompressive laminectomy so as to investigate the effect of HBO therapy on incomplete SCI in the plateau.

DETAILED DESCRIPTION:
History and current related studies Spinal cord injury (SCI) is a kind of serious disabling disease caused by various factors (such as trauma, infection), and can lead to paralysis. At present, 16-40 people/million suffer from SCI in developed countries every year; 34.3-60 people affect SCI in China every year. SCI is often caused by physical trauma, such as rotation, compression and hyperextension. This type of SCI is also known as traumatic spinal cord injury (TSCI). At present, there are many treatments for TSCI, but the prognosis is poor.

Hyperbaric oxygen (HBO) therapy is the medical use of oxygen at a level higher than atmospheric pressure for treating hypoxic disease (Hu et al., 2016). Secondary injuries, such as edema, neuronal necrosis, blood and spinal cord barrier disorders, have been shown to be strongly associated with a large number of inflammatory factors. HBO can effectively inhibit the generation of inflammatory factors, and promote repair and regeneration of neurons. Moreover, HBO can relieve hypoxia, protect the surrounding tissue, reduce the mitochondrial dysfunction in injury area, reduce bleeding area and reduce edema. HBO has been used to treat TSCI for a long time. Holbach et al. first found that HBO therapy improved postoperative dysfunction in TSCI patients. In recent years, a number of clinical studies have focused on HBO therapy for TSCI, and the patients recovered well. Atmospheric pressure is very low in the plateau, and oxygen content in plateau environment is less than that in plain area. Secondary apoptosis induced by ischemia and hypoxia after SCI is the main cause of spinal cord dysfunction. HBO therapy can increase the dissolved oxygen, which is helpful for the recovery of incomplete spinal nerve function. Therefore, HBO therapy has higher therapeutic value in plateau than in plain.

Data management The observation forms were filled out accurately, completely and timely by researchers. Data were recorded electronically by data managers using a double-data entry strategy. The electronic database was collated and locked only by the project manager. The locked electronic database could not be altered. All data regarding this trial were preserved by the Affiliated Hospital of Qinghai University, China. The electronic database was statistically analyzed by a professional statistician. Anonymized trial data will be published at www.figshare.com.

Statistical analysis Statistical analysis was performed using SPSS 22.0 software (IBM, Armonk, NY, USA). Measurement data were expressed as mean ± SD. Normality test and variance homogeneity test were conducted. Normally distributed data with homogeneity were compared using one-way analysis of variance. Non-normally distributed data were compared using Wilcoxon two-sample rank sum test. Ranked data were analyzed using rank sum test. A value of P < 0.05 was considered statistically significant. Results followed the intention-to-treat principle.

Confidentiality Identifying information, such as observation forms and informed consent, was password-protected and not altered for future reference. No person, other than an authorized researcher, may be in contact with it.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete spinal cord injury (SCI) (contusion) assessed by rectal examination in accordance with International standards for neurological classification of spinal cord injury (Revised 2011);
* SCI revealed by CT, X-ray or MRI scan;
* Clear trauma in the spine;
* Different degrees of movement, sensation and sphincter dysfunction below spine injury segment;
* Living in the plateau for at least 2 years;
* Age of ≥18 years, irrespective of sex.

Exclusion Criteria:

* Brain trauma, combined injury of chest and abdominal organs, instable vital signs or disturbance of consciousness;
* Coagulation dysfunction;
* Hypertension, heart disease, diabetes, stroke, brain damage and neurological disease;
* Lumbar surgery, trauma history, lumbar fracture, infection, tumor, severe osteoporosis;
* Nerve pain, limb cramps, periarticular heterotopic ossification;
* Other diseases that may impact neurological examination;
* Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Modified Barthel index | 40 days after treatment
  To assess the difference before and after treatment

SECONDARY OUTCOMES:
American Spinal Injury Association impairment scale grading | 40 days after treatment
  To assess the recovery of spine nerve function before and after treatment. American Spinal Injury Association(ASIA) is a spinal cord injury (SCI) neurological assessment criteria developed by the American Spinal Injury Association in 1982, contains grades A-E.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Ph.D, Principal Investigator — Affiliated Hospital of Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided